CLINICAL TRIAL: NCT05624346
Title: The Effect Of Respiratory Exercise After Laparoscopic Surgery On Pain, Anxiety, Nausea-Vomiting And Respiratory Parameters
Brief Title: The Effect of Respiratory Exercise After Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Suna Uzun, Student, Bartın Unıversity
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-SBB-0086
Record Dates: First submitted 2022-11-10; First posted 2022-11-22 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Laparoscopic Surgery; Breathing Exercise
Keywords: Laparoscopic Surgery; Breathing Exercise; Pain; Anxiety; Postoperative period
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental research
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): After the operation, breathing exercises will be applied to the patients.
  Interventions: Other: Deep-Breathing Exercises
- Control Group (No Intervention): There will be no intervention other than routine nursing care practices in the hospital.

INTERVENTIONS:
Other: Deep-Breathing Exercises — In addition to routine care in the hospital, the patient will be taught pre-operative breathing exercises. After surgery the patients do deep-breathing exercises every hour.
  Arms: Experimental Group

SUMMARY:
Laparoscopic surgery (LS) enables the patient to experience the desired result with smaller incisions in the postoperative period, more aesthetically, stress-free and less painful.

This increases patient satisfaction and reduces morbidity and mortality. In the literature, it has been stated that respiratory exercises reduce the level of anxiety in different patient groups in the postoperative period and increase the quality of sleep and recovery.

Among the duties and responsibilities of nurses working in surgical clinics are to provide breathing exercise training to patients in the preoperative period and to ensure that it is applied in the postoperative period.

This study was planned to determine the effect of respiratory exercise applied to laparoscopic surgery patients on postoperative pain, anxiety, nausea-vomiting and respiratory parameters.

DETAILED DESCRIPTION:
Surgical intervention is a form of treatment applied to preserve the physiology of the organism as much as possible, and to normalize the body functions that are impaired in diseases and injuries.

Laparoscopic surgery (LC) enables the patient to experience the desired result more aesthetically, stress-free and less painful with smaller incisions in the postoperative period. This increases patient satisfaction and reduces morbidity and mortality.

It is made with small incisions without exposing large tissues, which is inevitable in LC surgery. Less tissue dissection provides a lower level of neuroendocrine and metabolic response to stress in humans. Postoperative pain and need for analgesia are reduced. It accelerates the recovery process of the patient and helps him return to daily life in a shorter time. It reduces the patient's hospital stay. It increases comfort and quality of life, provides less suppression of the immune system.

LC has a lower mortality rate in addition to reducing the incidence of complications such as cosmetic problems, bleeding, injury, infection, inflammation, ileus. All these make LC more advantageous than other surgical methods. Pain, anxiety, nausea and vomiting are among the most common complications in the early postoperative period. In addition to pharmacological methods, non-pharmacological methods are also used to eliminate complications. Breathing exercise, which is the first step of relaxation, is one of the frequently used non-pharmacological methods.

With breathing exercises, it is ensured that the respiratory rate and depth are regulated, the muscles of the assisted respiration relax, and the efficiency of respiration is increased. The most commonly used breathing exercises are pursed lip breathing (pursed lip breathing) and diaphragmatic breathing. Nurses should explain the steps of the procedure in the exercise applications in a way that the patient can understand and ensure that they practice the exercises regularly.

Preoperative patient education, which can help prevent post-operative problems and early recovery; with explanation of surgical procedures, deep breathing, coughing, leg exercises, turning in bed, mobilization and reducing pain etc. includes topics. Among the duties and responsibilities of nurses working in surgical clinics are to provide breathing exercise training to patients in the preoperative period and to ensure its implementation in the postoperative period.

Post-operative patients are not ready to learn anything new due to pain and other reasons. Therefore, these trainings should be completed before the surgery. The purpose of giving deep breathing and coughing exercises; Expanding the decreased lung capacity during and after anesthesia, restoring the perfusion-ventilation balance and regulating its distribution, increasing oxygenation, protecting the airways, and enabling the secretions in the airways to be expelled more easily with effective coughing.

Teaching the breathing exercises, which is one of the basic duties of the surgical nurse, to the patients, explaining the importance of this and having it done regularly, increases the oxygenation of the tissues and affects the healing quality positively. In the literature, it has been stated that respiratory exercises reduce the level of anxiety and increase the quality of sleep and recovery in different patient groups in the postoperative period.

Nurses should take an active role in diagnosing nausea, vomiting, pain and respiratory problems that may occur in the postoperative period, planning and applying the necessary pharmacological and non-pharmacological methods, monitoring and evaluating the results of treatment, and should be able to prevent problems that may develop.

This study was planned to determine the effect of respiratory exercises on postoperative pain, anxiety, nausea-vomiting and respiratory parameters after laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study verbally and in writing,
* 18 years and over,
* No neurological or psychological problems,
* Fluent in Turkish and able to communicate,
* No respiratory disease,
* Brought to the post-operative service,
* Planned cases,
* Patients who underwent laparoscopic general surgery (such as laparoscopic cholecystectomy, colon, inguinal hernia, appendectomy, incisional hernia, sleeve gastrectomy) under general anesthesia were included in the study.

Exclusion Criteria:

* Those who do not accept to participate in the study verbally or in writing,
* Not 18 years of age or older
* Having neurological or psychological problems,
* Those who do not speak Turkish and cannot communicate
* Having respiratory disease
* Transferred to the intensive care unit after surgery,
* Emergency and unplanned cases
* Cases that converted from laparoscopic surgery to open surgery under general anesthesia were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Measuring of anxiety | Between 1-6 hours and 24 hours after surgery
  The effect of breathing exercise in patients after laparoscopic surgery using by State and Trait Anxiety Scale. The State-Trait Anxiety Inventory is one of the first tests to assess both state and trait anxiety separately. Each type of anxiety has its own scale of 20 different questions that are scored. Scores range from 20 to 80, with higher scores correlating with greater anxiety.

SECONDARY OUTCOMES:
Respiratory parameters | 2nd, 6th, 12th and 24th hours after surgery
  The effect of deep breathing exercises on respiratory parameters in patients with laparoscopic surgery using a saturation device.
Measuring the level of nausea-vomiting | 2nd, 4th, 6th, 12th and 24th hours after surgery
  The effect of deep breathing exercises on nausea-vomiting in patients with laparoscopic surgery using by nausea severity scale.
Measuring the level of pain | 2nd, 6th, 12th and 24th hours after surgery
  The effect of deep breathing exercises on pain in patients with laparoscopic surgery using by Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Suna UZUN, Msc. Student, Principal Investigator — Bartın Unıversity; Elif KARAHAN, Assoc. Prof., Study Director — Bartın Unıversity
Locations (1):
- Bartin Hospital of State, Bartın, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT05624346/Prot_000.pdf